CLINICAL TRIAL: NCT06834087
Title: Comparative Evaluation of Methylene Blue and Methylene Blue Nanoparticles Assisted Photodynamic Therapy As Adjunctive to Laser Treatment of Physiological Gingival Pigmentation: a Randomized Controlled Clinical Trial
Brief Title: Laser Treatment with Methylene Blue Vs. Nanoparticle-Assisted Photodynamic Therapy for Gingival Pigmentation: a Randomized Clinical Trial
Acronym: MB-Laser-GP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Roaa Hadi Hussein Jasem (Other)
Responsible Party: Sponsor-Investigator, Roaa Hadi Hussein Jasem, B.D.S. 2013 ALANBAR UNIVERSITY FACULTY OF DENTISTRY, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kfsirb200-489
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Physiological Gingival Pigmentation
Keywords: Gingival Pigmentation, Laser Therapy, Photodynamic Therapy, Methylene Blue, Nanoparticles, Periodontology, Aesthetic Dentistry
MeSH Terms: interventions — Photochemotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (Control Group) Laser-Only Treatment (Other): Patients in this group will undergo laser-assisted gingival depigmentation using a diode laser (970 nm wavelength, 2.0 W power, continuous mode) with a 200 µm fiber tip applied for 30 seconds per site in contact mode.
  Interventions: Procedure: Laser-Assisted Gingival Depigmentation
- Arm 2 (Experimental Group 1) PDT with Conventional Methylene Blue + Laser (Experimental): This group will receive photodynamic therapy (PDT) using a conventional methylene blue solution (0.1%), applied for 2 minutes before activation with a 660 nm diode laser (1.5 W, pulsed mode, 60 seconds per site). This will be followed by laser-assisted gingival depigmentation using a diode laser (970 nm wavelength, 2.0 W power, continuous mode, 200 µm fiber tip, 30 seconds per site).
  Interventions: Drug: Photodynamic Therapy with Conventional Methylene Blue
- Arm 3 (Experimental Group 2) PDT with Methylene Blue Nanoparticles + Laser (Active Comparator): Patients in this group will receive PDT with methylene blue nanoparticles (0.1%) applied for 2 minutes before activation with a 660 nm diode laser (1.5 W, pulsed mode, 60 seconds per site). This will be followed by laser-assisted gingival depigmentation using a diode laser (970 nm wavelength, 2.0 W power, continuous mode, 200 µm fiber tip, 30 seconds per site).
  Interventions: Drug: Photodynamic Therapy with Methylene Blue Nanoparticles

INTERVENTIONS:
Procedure: Laser-Assisted Gingival Depigmentation — This intervention involves the use of a diode laser (970 nm wavelength, 2.0 W power, continuous mode) with a 200 µm fiber tip. The laser is applied in a sweeping motion over the pigmented gingiva in contact mode for 30 seconds per site to achieve depigmentation.
  Arms: Arm 1 (Control Group) Laser-Only Treatment
Drug: Photodynamic Therapy with Conventional Methylene Blue — This intervention consists of applying a 0.1% methylene blue solution to the pigmented gingiva for 2 minutes before activation with a diode laser (660 nm wavelength, 1.5 W power, pulsed mode) for 60 seconds per site. This is followed by laser-assisted gingival depigmentation using a 970 nm diode laser (2.0 W, continuous mode, 200 µm fiber tip, 30 seconds per site).
  Arms: Arm 2 (Experimental Group 1) PDT with Conventional Methylene Blue + Laser
Drug: Photodynamic Therapy with Methylene Blue Nanoparticles — This intervention involves the application of 0.1% methylene blue nanoparticles to the pigmented gingiva for 2 minutes to allow deeper tissue penetration. It is then activated using a diode laser (660 nm wavelength, 1.5 W power, pulsed mode) for 60 seconds per site, followed by laser-assisted gingival depigmentation using a 970 nm diode laser (2.0 W, continuous mode, 200 µm fiber tip, 30 seconds per site).
  Arms: Arm 3 (Experimental Group 2) PDT with Methylene Blue Nanoparticles + Laser

SUMMARY:
This randomized controlled clinical trial aims to compare the effectiveness of methylene blue and methylene blue nanoparticles as adjuncts to photodynamic therapy in laser treatment of physiological gingival pigmentation. The study evaluates pigmentation reduction, recurrence rates, healing time, and patient satisfaction. Conducted at Kafrelsheikh University, it includes three patient groups: laser-only treatment, conventional methylene blue-assisted PDT with laser, and methylene blue nanoparticles-assisted PDT with laser. The findings will contribute to advancements in aesthetic dentistry and laser-assisted depigmentation techniques.

ELIGIBILITY:
Inclusion Criteria:

Patients with physiological gingival pigmentation confirmed by clinical examination.

Age range: 18-50 years.

Patients with no history of systemic diseases or conditions that could affect wound healing (e.g., diabetes, autoimmune diseases).

Patients willing to undergo laser treatment and provide informed consent.

Non-smokers or individuals who have stopped smoking for at least six months.

Exclusion Criteria:

Patients with pathological gingival pigmentation (e.g., associated with syndromes or systemic conditions).

Use of medications affecting pigmentation or healing (e.g., anticoagulants, immunosuppressants).

Pregnant or lactating women or those taking contraceptive drugs.

Individuals with known allergies to methylene blue or nanoparticles.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-09-14 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Reduction in Gingival Pigmentation | Baseline, 1 Month, 3 Months, and 6 Months Post-Treatment
  The primary outcome will be assessed by evaluating changes in gingival pigmentation using clinical photographs and a standardized pigmentation index. Digital images of the treated gingival areas will be analyzed for pigmentation intensity reduction using imaging software. The pigmentation index scores range from:
  Score 0: Absence of pigmentation
  Score 1: Spots of brown to black color
  Score 2: Brown to black patches without diffuse pigmentation
  Score 3: Diffuse brown to black pigmentation

SECONDARY OUTCOMES:
Healing Time | 1 Month Post-Treatment
  The duration required for complete epithelialization of the treated gingival area will be recorded. Visual inspection at follow-up visits will determine the time until there is no visible inflammation, erythema, or delayed healing.
Patient Satisfaction | 1 Month, 3 Months, and 6 Months Post-Treatment
  Patient satisfaction will be assessed using a Visual Analog Scale (VAS) questionnaire. Patients will rate their satisfaction with the treatment, including aesthetic improvement, comfort during the procedure, and overall experience on a scale from 0 (completely dissatisfied) to 10 (completely satisfied).
Recurrence of Gingival Pigmentation | 3 Months and 6 Months Post-Treatment
  The degree of gingival pigmentation recurrence will be evaluated using clinical and photographic records. Re-pigmentation percentage will be calculated and documented at each follow-up visit.
Adverse Events | Throughout the study duration (up to 6 Months Post-Treatment)
  Any adverse effects such as persistent erythema, ulceration, or patient-reported pain post-treatment will be documented. A scoring system will be used to assess the severity of these events (e.g., mild, moderate, severe).

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Faculty of Oral and Dental Medicine, Kafr ash Shaykh, Kafr Ash Shaikh/ Elhamrawy, Egypt